CLINICAL TRIAL: NCT00224965
Title: Early Tobacco Abstinence in High Risk Smokers
Brief Title: Early Tobacco Abstinence - 5
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NIDA-13334-5; P50-13334-5
Record Dates: First submitted 2005-09-22; First posted 2005-09-23 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2005-09

CONDITIONS: Tobacco Use
Keywords: nicotine dependence
MeSH Terms: conditions — Tobacco Use; Tobacco Use Disorder | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
This proposal will conduct a prospective examination of the clinical course (intensity, content and duration) of tobacco (nicotine) abstinence effects in male and female smokers who are either heavy/light alcohol drinkers with/without depressive symptoms.

DETAILED DESCRIPTION:
1. To compare male and female smokers, with and without current depressive symptoms, in a prospective study of the intensity, content & duration of nicotine abstinence effects during an eight-day abstinence period, and responses to cue exposure (invivo cigarette cues, alcohol and negative affect-inducing imagery cues) during acute vs. prolonged abstinence and,
2. To compare male and female smokers, who are either heavy alcohol drinkers or light alcohol drinkers, in a prospective study of the intensity, content & duration of nicotine abstinence effects during an eight-day abstinence period, and responses to cue exposure (invivo cigarette cues, alcohol and negative affect-inducing imagery cues) during acute vs. prolonged abstinence.

ELIGIBILITY:
Inclusion Criteria:

1) between ages 18-60 years; (2) able to read and write English (3) SMOKER: Smoking >10 cigarettes per day for at least 1 year, with CO > 10 ppm, and blood cotinine concentration of 150 ng/ml or greater, FTND scores > 5.

(4) DEPRESSED SUBJECT: Not meeting SCID criteria for current major depression or more than one past major depressive episode, but having scores > 10 on the CES-D indicating presence of depressive symptomatology (5) NON-DEPRESSED SUBJECT: Not meeting SCID criteria for current major depression or more than one past major depressive episode, CES-D scores <10.

(6) HEAVY DRINKER: Not meeting SCID criteria for current alcohol dependence; drinking 20 or more drinks per month.

(7) LIGHT DRINKER: Not meeting SCID criteria for current alcohol dependence; drinking ten drinks or less per month

Exclusion Criteria:

1. Current dependence on cocaine, marijuana, opiates or alcohol
2. Positive urine screen for marijuana, cocaine or opiates at any appointment after the intake appointment.
3. Regular use of any psychoactive drugs including anxiolytics and antidepressants;
4. Current major depression or other psychiatric conditions
5. Subjects with any significant, untreated current medical conditions condition such as neurological, endocrine, cardiovascular, renal, liver, thyroid pathology or on medications for any recent medical events 6) Pregnant or lactating women -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140
Dates: Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie O'Malley, Ph.D., Principal Investigator — Substance Abuse Treatment Unit
Locations (1):
- Yale University, Dept. of Psychiatry, Minneapolis, Minnesota, United States